CLINICAL TRIAL: NCT06074991
Title: The Effect of Music Therapy on Pain and Anxiety in Intensive Care Patients
Brief Title: The Effect of Music Therapy on Pain and Anxiety
Acronym: AtaturkU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: Nurse Researcher Fatih BÜDÜŞ (Unknown)
Responsible Party: Principal Investigator, Kübra Gökalp, Phd, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2023
Record Dates: First submitted 2023-04-05; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pain; Anxiety; Music-Induced Seizure
Keywords: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Music therapy was applied to the patients in the experimental group with the help of mp3 and headphones for 30 minutes in a position where they felt comfortable. Hüseyni makam was used for music therapy. Posttest-1 data were collected immediately after the end of the music therapy. 30 minutes after the posttest-1 data, the posttest-2 data were collected. The patients in the control group, on the other hand, did not undergo any procedure other than medical intervention. Posttest-1 data were collected 30 minutes after the pretest and posttest-2 data 30 minutes after the posttest-1.
  Interventions: Other: musıc therapy
- control group (No Intervention): The control group did not receive any therapy, and there was no interaction between the experimental group and the control group during the training period.

INTERVENTIONS:
Other: musıc therapy — Music therapy was applied to the patients in the experimental group with the help of mp3 and headphones for 30 minutes in a position where they felt comfortable. Hüseyni makam was used for music therapy.
  Arms: experimental group

SUMMARY:
This study will be conducted to determine the effect of music therapy on pain and anxiety following coronary angiography in patients in intensive care. 60 patients who underwent coronary angiography will be randomized and divided into experimental (n = 30) and control (n = 30) groups. "Personal Data Form", "Pain Visual Analog Scale (Pain-VAS)", "Anxiety Visual Analog Scale (Anxiety-VAS)" and "Richmond Agitation and Sedation Scale (RASS)" were used to collect data. While participants in the experimental group will be given a problem-solving training program, no intervention will be made to the control group. The data in the control and experimental groups will be distributed homogeneously.

DETAILED DESCRIPTION:
Personal Data Form The form, which was prepared by the researchers by scanning the literature, consists of questions questioning the patients' age, gender, marital status, socioeconomic status, the post-operative day, whether they had previous intensive care experience, whether they had a psychiatric diagnosis, and the Glasgow Coma Scale score.

Pain Visual Analog Scale Pain-VAS, the validity and reliability of which was tested by Price, McGrath, Rafii, and Buckingham58, is a measurement tool that measures both pain intensity and pain relief, which is easy, effective, repetitive and requires minimal tools. It is a one-dimensional scale whose validity and reliability studies have been carried out in Turkey and which is used to measure subjective components of pain intensity. The VAS is a 10 cm long ruler drawn horizontally or vertically, starting with "No pain" and ending with "Unbearable pain".

Anxiety Visual Analog Scale Although the use of the visual analogue scale dates back to the early 20th century, its worldwide use became widespread in 1969 with the research of Zealley and Aitken.60 The VAS typically consists of a 10-centimeter closed-end line. At either end of this line are words describing the two extremes of the emotion to be measured (for example, Zero-Maximum). Patients are asked to mark where their current feeling is anywhere on the scale, and the distance from the minimum (zero) end gives the patient's score.

Richmond Agitation and Sedation Scale RASS was developed in collaboration with a multidisciplinary team at the University of Virginia as a result of studies at Richmond Virginia Commonwealth University. 61 Turkish Validity and Reliability Study was conducted by Sılay and Akyol62. RASS is a 10-stage scoring system in which patients are evaluated by making eye contact apart from verbal stimuli. Although there are many scales used to evaluate patients in intensive care units with adult patients, the RASS has a very good rating compared to these scales. RASS scale is evaluated between -5 level and +4 level. As it decreases to -5 level, the patient's sedation increases, and as it rises to +4 level, his agitation increases. Our most ideal level is 0.

Research data will be collected by the researcher using face-to-face interview technique.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study voluntarily,
* Being open to communication,
* be over 18 years old,
* Application of coronary angiography for the first time,
* Having a score of 0 or higher according to the Ramsay Sedation Scale,
* Being on the first day of intensive care treatment,
* This is the first time he is being treated in the intensive care unit.

Exclusion Criteria:

* By-pass decision after coronary angiography,
* Transferring the patient to the ward after coronary angiography,
* Having additional psychiatric disorders,
* Being hospitalized in intensive care before,
* It is the presence of delirium in the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | 0,30,60 minutes
  Pain-VAS, the validity and reliability of which was tested by Price, McGrath, Rafii, and Buckingham, is a measurement tool that measures both pain intensity and pain relief, which is easy, effective, repetitive and requires minimal tools. It is a one-dimensional scale whose validity and reliability studies have been conducted in Turkey and which is used to measure subjective components of pain intensity. VAS is 10 cm long drawn horizontally or vertically. It is a ruler that starts with 0cm "No pain" and ends with 10cm "Unbearable pain".Change from Pain-VAS at 60 minutes.
Anxiety Visual Analog Scale | 0,30,60 minutes
  Although the beginning of the use of the visual analog scale dates back to the early 20th century, its worldwide use became widespread in 1969 with the research of Zealley and Aitken. The VAS typically consists of a 10-centimeter double-ended line. At either end of this line are words describing the two extremes of the emotion to be measured (for example, Zero-Maximum). Patients are asked to mark where their current feeling is anywhere on the scale, and the distance from the minimum (zero) end gives the patient's score.Change from Anxiety-VAS at 60 minutes.

SECONDARY OUTCOMES:
Richmond Agitation and Sedation Scale | 0,30,60 minutes
  RASS was developed in collaboration with a multidisciplinary team at the University of Virginia as a result of studies at Richmond Virginia Commonwealth University. Turkish Validity and Reliability Study was conducted by Sılay and Akyol. RASS is a 10-stage scoring system in which patients are evaluated by making eye contact apart from verbal stimuli. RASS scale is evaluated between -5 level and +4 level. As it decreases to -5 level, the patient's sedation increases, and as it rises to +4 level, his agitation increases. Our most ideal level is 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No